CLINICAL TRIAL: NCT01422356
Title: Human Papillomavirus (HPV) Infection in Young Men Who Have Sex With Men
Acronym: HYPER
Status: Completed | Type: Observational
Sponsor: The Alfred (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Christopher Fairley, Professor of Public Health Central Clinical School Monash University and Director Melbourne Sexual Health Centre Alfred Health, The Alfred
Other Study IDs: MSHC-174/10
Record Dates: First submitted 2011-08-16; First posted 2011-08-24 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2013-12

CONDITIONS: Human Papillomavirus
Keywords: cohort study; men who have sex with men
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genital samples (genital swabs from anus, penis), oral rinse, and serum.
Oversight: Data Monitoring Committee: No

SUMMARY:
Studies indicate that men who have sex with men (MSM) have a high prevalence of anogenital Human papillomavirus (HPV) infection and increased risk for HPV related anogenital lesions including anogenital warts, anal intraepithelial neoplasia (the abnormal proliferation of cells) and anal cancer. Currently in Australia, HPV vaccine for men is not covered by programs. This study will explore the prevalence of HPV infection and sexual behaviours associated with varying prevalence of HPV infection.

The investigators will survey 200 MSM aged 16-20 years who just started their sexual life. The investigators will use a questionnaire to collect information of socio-demographic characteristics, lifetime sexual experience, recent sexual experience, the most recent sexual contact, sexually transmitted infections (STIs)/HIV history and testing history, HPV knowledge and attitude, smoking/alcohol/drug/circumcision. The investigators will also collect oral, penile and anal samples as well as blood samples to test for HPV DNA and antibody.

The study will include four visits in the 12-month period. In each visit, participants will be asked to fill a questionnaire and provide oral, penile and anal samples as well as blood samples.

DETAILED DESCRIPTION:
Study aims

The objectives of this study are to determine among younger MSM:

1. The prevalence of HPV infection
2. Sexual behaviours associated with varying prevalence of HPV infection

Methods

Criteria for eligibility:

* Men aged 16 to 20
* Same sex attracted
* Able to complete all study requirements including questionnaire in English and completion of 4 visits

Recruitment

Men were recruited between October 2010 and September 2012 via a number of avenues focusing on gay teenage males: community organizations supporting gay teenagers with study promotion at social events such as dance parties; gay clubs at six Melbourne universities; gay community events including the MidSumma Festival; gay media including radio and magazine; the study website; and social networking websites including Facebook, Twitter and Grindr. Recruitment also took place through three sexual health services in Melbourne.

Men were assessed by the study nurse at a baseline visit then 3, 6, and 12 months later. On each occasion specimens were obtained for HPV DNA testing, blood was obtained for HPV serology, and men completed a questionnaire regarding their sexual experiences.

Specimen collection Specimens were obtained from men for HPV DNA testing in the following order: first an oral rinse, second an anal canal swab, third a perianal swab, then fourth a penile swab. The oral rinse and penile swab were self-collected by men after watching a video demonstrating how to self-collect these specimens

Men were screened for pharyngeal and rectal Neisseria gonorrhoeae using modified Thayer-martin media. First void urine and a rectal swab were tested for Chlamydia trachomatis by strand displacement assay (Becton Dickinson ProbeTec ET, NJ, USA). In addition, men were screened for syphilis using enzyme immunoassay (EIA) and rapid plasma reagin and tested for HIV using EIA.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 16 to 20
* Same sex attracted
* Able to complete all study requirements including questionnaire in English and completion of 4 visits

Ages: 16 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Young same sex attracted men 16-20 years of age from Melbourne
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher K Fairley, MB BS, Ph D, Principal Investigator — The Alfred
Locations (1):
- Alfred Health (Melbourne Sexual Health Centre), Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Chow EPF, Fairley CK, Zou H, Wigan R, Garland SM, Cornall AM, Atchison S, Tabrizi SN, Chen MY. Human Papillomavirus Antibody Levels Following Vaccination or Natural Infection Among Young Men Who Have Sex With Men. Clin Infect Dis. 2022 Aug 25;75(2):323-329. doi: 10.1093/cid/ciab1052. PMID 34971362
- [Derived] Chow EPF, Tabrizi SN, Fairley CK, Wigan R, Machalek DA, Garland SM, Cornall AM, Atchison S, Hocking JS, Bradshaw CS, Balgovind P, Murray GL, Chen MY. Prevalence of human papillomavirus in young men who have sex with men after the implementation of gender-neutral HPV vaccination: a repeated cross-sectional study. Lancet Infect Dis. 2021 Oct;21(10):1448-1457. doi: 10.1016/S1473-3099(20)30687-3. Epub 2021 May 24. PMID 34043963
- [Derived] Zou H, Tabrizi SN, Grulich AE, Hocking JS, Bradshaw CS, Cornall AM, Morrow A, Prestage G, Law MG, Garland SM, Chen MY, Fairley CK. Site-specific human papillomavirus infection in adolescent men who have sex with men (HYPER): an observational cohort study. Lancet Infect Dis. 2015 Jan;15(1):65-73. doi: 10.1016/S1473-3099(14)70994-6. Epub 2014 Nov 28. PMID 25435055

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two hundred males aged 16 to 20 years were recruited into the study. Men were seen at 0, 3, 6 and 12 months.
Groups:
- 12 Month Cohort: 16-20 year old males
Period: Overall Study
Arm/Group | 12 Month Cohort
Started | 200
Completed | 169
Not Completed | 31

BASELINE CHARACTERISTICS:
Arm/Group | 12 Month Cohort
Number analyzed (Participants) | 200
Age, Continuous [Median (Full Range); unit: years] | 19 [16 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 200
Region of Enrollment [Number; unit: participants]
  Australia | 200

OUTCOME MEASURES:

1. Primary Outcome: HPV Prevalence
Description: Prevalence of anal HPV of any type at baseline
Time Frame: Baseline
Population: Number of men at baseline visit
Measure: Number; unit: participants
Arm/Group | Baseline Prevalence
Number analyzed (Participants) | 200
participants | 61

ADVERSE EVENTS:
Arm/Group | 12 Month Cohort
Serious Adverse Events (participants affected / at risk) | 0/200
Other Adverse Events (participants affected / at risk) | 0/200

LIMITATIONS AND CAVEATS:
The findings from this study may or may not extend to other populations of teenage MSM.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less